CLINICAL TRIAL: NCT02527330
Title: Evaluation of Myocardial Iron Deposition in Patients of Heart Failure Using T2* MR Imaging
Acronym: CHFIRONMR
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-2770A3
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2016-08

CONDITIONS: Heart Failure; Iron Overload; Cardiomyopathies
Keywords: Myocardial iron deposition; T2* imaging; heart failure
MeSH Terms: conditions — Heart Failure; Iron Overload; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control group: Age- and gender-matched healthy volunteers recruited as normal control group.
  Interventions: Other: MR T2* imaging
- Stable HF group: Patients with acute HF episode with hospitalization treatment within 12 months, LVEF>=55%
  Interventions: Other: MR T2* imaging
- Unstable HF group: Patients with acute HF episode with hospitalization treatment within 12 months, currently LVEF<55%.
  Interventions: Other: MR T2* imaging

INTERVENTIONS:
Other: MR T2* imaging — Cardiac magnetic resonance imaging with T2* imaging

SUMMARY:
Heart failure from myocardial iron deposition is a severe complication for patients with hematological disorders who need repeated blood transfusions. Increased cardiac iron content impacts the contractility of cardiomyocytes and can also lead to myocarditis, pericarditis, and arrhythmias. The severity of cardiac dysfunction depends on the amount of iron deposited in the myocardium.

Cardiovascular magnetic resonance (CMR) imaging is used as noninvasive method to evaluate the amount of iron in the heart. Myocardial T2* value has been shown to correlate well with biopsy-derived iron concentration in the heart, and myocardial T2* values less than 20ms (indicating elevated iron) were found to be associated with LV dysfunction and improve in concert with LV function during recovery. The majority of the recent studies about myocardial iron overload and the effect of iron chelation therapy were focused on patients with transfusion-dependent hematological disorder, especially beta-thalassemia major.

The objective of this 3-year project is to evaluate myocardial iron deposition in patients with heart failure, induced by variable causes. With myocardial T2* imaging, the investigators will analyze the decreased signal intensity in the ventricular septum and quantitatively acquire the T2* value as marker for myocardial iron deposition. The first year is a cross-sectional study. The investigators aim to compare the severity of myocardial iron deposition of normal subjects and that of stable HF patients in recovery with normal or impaired ejection fraction (EF). Total 60 subjects will be enrolled, with 20 subjects in each group. In the 2nd and 3rd years, the investigators plan a prospective longitudinal study of 40 subjects. Enrolled patients will be evaluated with cardiac T2* imaging at three time points, i.e., disease onset, 6 months and one year after treatment, and will be followed up until the end of this project (1.5~3-year follow up). In total 120 MR scans will be performed in the 2nd and 3rd years. The presence and severity of myocardial iron deposition will be correlated with the disease course, patient biochemistry data and clinical outcome.

DETAILED DESCRIPTION:
Introduction

Heart failure (HF) is a complex clinical syndrome resulting from any structural or functional cardiac disorder that impairs the ability of the ventricle to fill with or eject blood. In Taiwan, HF is a growing epidemic, owing to the aging population and the increasing survival of patients presenting with acute myocardial infarction and various other heart diseases. The reported 5- and 10-year mortality ranged from 14% and 48.2% in those with impaired LVEF versus 14.1% and 24.4% in those with pre- served LVEF, respectively.

The diagnosis of HF is based on symptoms typical of heart failure, and signs typical of heart failure and an objective evidence structural or functional abnormality of the heart. Asymptomatic structural or functional abnormalities of the heart (myocardial remodeling) are usually progressive disorders and are considered as precursors of symptomatic heart failure. Therefore early diagnosis of the underlying etiology and cause should always be sought for guiding a suitable and preventive treatment.

Myocardial iron deposition leads to progressive heart dysfunction and is thought to be a leading cause of death in transfusion-dependent anemia. Endomyocardial biopsy, which has been used to evaluate iron deposition in the heart, is risky and has unacceptable sampling variability. Non-invasive MR scanning is currently the imaging method shown to be reliable and accurate to assess myocardial iron loading. The application of the MR transverse relaxation times T2* has been successfully demonstrated for quantitative assessment of the iron concentration in the heart.

Purpose The objective of this project is to evaluate myocardial iron deposition in patients with heart failure (HF). Deposition of iron on the myocardium is expected to be found in patients with heart failure induced by other cause rather than transfusion-dependent hematological disorder. In this longitudinal study, we will attempt to analyze the presence and severity of myocardial iron deposition, variation along the course and correlate with clinical outcome in patients with HF.

Methods This is a 3-year project on human subjects focusing on myocardial iron deposition. Direct myocardial iron measurement using endomyocardial biopsy is risky and has unacceptable sampling variability. Therefore MR T2* imaging is chosen in this project due to non-invasiveness and T2* value quantitatively correlates with the severity of myocardial iron overload.

The inclusion criteria for this study are: (1) heart failure patients diagnosed in the Keelung Chang Gung Memorial Hospital; (2) patients must be ≥ 20 and ≤ 70 years of age; (3) patients must be willing to undergo standard treatment and follow up in the Heart Failure Center; (4) patients must be able to give informed consent. The exclusion criteria are: (1) patients who are judged to be noncompliant to treatment or not accessible for follow up; (2) patients with contraindications to MR scanning, such as claustrophobia, cardiac pacemaker, metal implants, or unable to cooperate for MRI study due to mental status; (3) Severe renal function impairment (glomerular filtration rate less than 30 mL/min/1.73m2); (4) pregnant or breast-feeding; (5) history of open-heart surgery. Medical records of eligible patients will be identified and centrally reviewed in the project joint meeting before enrollment to ensure the study quality.

1. st year plan The first year is a cross-sectional study. By using T2* imaging, we aim to compare the severity of myocardial iron deposition of normal subjects and that of stable HF patients in recovery with normal or impaired ejection fraction (EF). Total 60 subjects will be enrolled, with a group of treated HF patients with normal EF (n=20), a group of treated HF patients with impaired EF (n=20), and a control group (n=20). The control group consists of age and gender matched normal volunteers without previously documented cardiac disease. In this part, to compare the T2*value of the HF patient group and the normal group, two-sample t equality test will be considered and sample size can be chosen to achieve an 80% power for detecting a clinically meaningful difference at level of significance α=0.05. The G*Power 3.1.4 software 4 is utilized to compute required sample size for the first year study. The two-independent-sample t-test with the effect size of 0.74, level of significance α=0.05, and power of 0.8 requires a total sample of 60 participants (20 for each group). The clinically meaningful effect size is set at 0.74 according to our small pilot studies.
2. nd and 3rd years In the 2nd and 3rd years, we plan a prospective longitudinal study of 40 subjects. Enrolled patients will be evaluated with cardiac MR T2* imaging at three time points, i.e., disease onset, 6 months and one year after treatment, and will be followed up until the end of this project (1.5~3-year follow up). Therefore in total 120 MR scans will be performed in the 2nd and 3rd years. The presence and severity of myocardial iron deposition will be correlated with the disease course, patient biochemistry data and clinical outcome.

MRI imaging and data analysis

Cardiac MRI will be performed in a 3-T MRI scanner with intravenous administration of gadolinium-based MR contrast medium for the HF subjects, in order to identify any ischemia foucs and assess myocardial viability. For all the test subjects, EF will be calculated with Simpson disk summation method using short-axis cine steady-state free precession images of the left ventricle (LV) as previously reported (12). LV endocardial borders will be semi-automated traced on each short-axis image obtained in both end-diastole and end-systole to determine the ventricular cavity area for each slice. The area of the tracing for each image slice will be multiplied by the slice interval (slice thickness plus image gap) to determine a volume for that slice. The volumes of the slices will be summed to determine an LV volume. LVEF can be determined by end-diastolic volume (EDV) and end-systolic volume (ESV) using the following equation:

LVEF = stroke volume (EDV - ESV) ÷ EDV ………………………………………………. (1)

Iron in the myocardium was quantified by measuring T2* (1/R2*), a MR relaxation parameter that has been shown to vary inversely with tissue iron concentration. This technique has high reproducibility and inter-MRI scanner agreement. MRI measurements will be performed using a 3-T clinical MRI scanner (Skyra, Siemens AG) with a new pulse sequence (Multi Echo GRE, WIP 732, Siemens). Myocardial T2* will be assessed with the use of a single breath-hold multiecho technique. In brief, a single 10-mm-thick short-axis mid-ventricular slice of the LV will be acquired at 8 echo times with standard shimming in a single breath-hold. For analysis, a full-thickness region of interest will be chosen in the interventricular septum. The signal intensity of this region will be measured for each image with the use of in-house designed software (CMRtools, Cardiovascular Imaging Solutions, London, UK).

Statistical analysis plan Descriptive statistics will be calculated for all characteristics of the study subjects. For continuous data, two-independent-sample t-test will be used to test the difference of T2* value between two groups, and methods of analysis of variance (ANOVA) will be used to assess difference between 3 or more groups. The non-parametric methods of Mann-Whitney U or Kruskal-Wallis H will be used to compare two or more groups for small sample size or continuous variables not following the normal distribution. The Pearson's chi-square test will be used to evaluate the association between variables. The Spearman's rho test will be used to correlate LVEF and T2* value measured by MRI.

Expected problems and difficulties

One of the large hurdles to overcome is patient collection because this project involves clinical imaging and follow up. For the close coordination of researchers in various departments and good operation of the patients, we need an in-house research assistant to assure the workflow and data completeness.

Because T2* at high field decreases substantially and its quantitation is vulnerable to increased B0 inhomogeneity, it is especially challenging at 3T. Therefore we will integrate a committed, interdisciplinary team of radiologist, and MR physicists to overcome these challenges.

To solve the technical challenges accompanied with the high field strength 3 Tesla systems such as field inhomogenicity and susceptibility artifact. Second-order shimming (water peak line width, 4.7 Hz) has been proven in 3 Tesla MR system to be better than first-order (16.5 Hz) and iterative shimming (18 Hz) and will be applied in this project to improve the correction of air and tissue susceptibility differences.

Use of instruments The MR T2* imaging study will be performed in a 3-Tesla Siemens Skyra MR system at Keelung Chang Gung Memorial Hospital. There will be 60 scans in the 1st year, and 120 scans in the 2nd and 3rd years. In total 180 MR scans will be arranged over 3 years. Given 45 working weeks per year, on average there will be 1.3 scan per week. Each cardiac MR study will require 2 scan slots (about 2 hours) plus post-processing time, and will be charged as only one slot. The scanner time occupancy is approved under the MRI regulation of Department of Radiology.

ELIGIBILITY:
Inclusion Criteria:

1. heart failure patients diagnosed in the Keelung Chang Gung Memorial Hospital
2. patients must be ≥ 20 and ≤ 70 years of age
3. patients must be willing to undergo standard treatment and follow up in the Heart Failure Center
4. patients must be able to give informed consent.

Exclusion Criteria:

1. patients who are judged to be noncompliant to treatment or not accessible for follow up
2. patients with contraindications to MR scanning, such as claustrophobia, cardiac pacemaker, metal implants, or unable to cooperate for MRI study due to mental status
3. Severe renal function impairment (glomerular filtration rate less than 30 mL/min/1.73m2)
4. pregnant or breast-feeding
5. history of open-heart surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute HF episode with hospitalization treatment within 12 months were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
T2* Values | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan